CLINICAL TRIAL: NCT06592482
Title: A Phase I, Single-Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD0780
Brief Title: A Phase I Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD0780
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7960C00007
Record Dates: First submitted 2024-06-12; First posted 2024-09-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: AZD0780 (Experimental): Participants with severe renal impairment (eGFR < 30 mL/min), not on dialysis.
  Interventions: Drug: AZD0780
- Group 2: AZD0780 (Experimental): Participants with ESRD (eGFR < 15 mL/min) on a stable intermittent HD schedule for at least 3 months prior to planned dosing.
  Interventions: Drug: AZD0780
- Group 3: AZD0780 (Experimental): Participants with normal renal function demographically matched by sex, age, and body mass index (BMI) to the impaired participants (eGFR of ≥ 90 mL/min)
  Interventions: Drug: AZD0780
- Group 4 (optional): AZD0780 (Experimental): Participants with moderate renal impairment (eGFR ≥ 30 to < 60 mL/min).
  Interventions: Drug: AZD0780

INTERVENTIONS:
Drug: AZD0780 — A single "A" dose of AZD0780 will be administered in the morning on Day 1 under fasted condition. Study intervention will be administered orally with approximately 240 mL of water.

SUMMARY:
This is a Phase I, multi-centre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD0780 in male and female participants (females of non-childbearing potential) with severe renal impairment not on dialysis, end-stage renal disease (ESRD) on intermittent haemodialysis (HD), or moderate renal impairment (optional) compared with male and female participants (females of non-childbearing potential) with normal renal function. Potential participants will be screened to assess their eligibility to enter the study up to 4 weeks prior to administration of study intervention. Eligible participants will be admitted to the study site on Day -1. On Day 1, an "A" single oral dose of AZD0780 will be administered, and participants will be confined to the study site until after assessments are completed on Day 11.

DETAILED DESCRIPTION:
This is a Phase I, multi-centre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD0780 in male and female participants (females of non-childbearing potential) with severe renal impairment not on dialysis, end-stage renal disease (ESRD) on intermittent haemodialysis (HD), or moderate renal impairment (optional) compared with male and female participants (females of non-childbearing potential) with normal renal function.

Participants will be assigned to the following groups based on body surface area-adjusted estimated glomerular filtration rate (eGFR) determined by a local laboratory at screening by the Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation (2021) using serum creatinine:

Group 1: Participants with severe renal impairment (eGFR < 30 mL/min), not on dialysis.

Group 2: Participants with ESRD (eGFR < 15 mL/min) on a stable intermittent HD schedule for at least 3 months prior to planned dosing.

Group 3: Participants with normal renal function demographically matched by sex,age, and body mass index (BMI) to the impaired participants (eGFR of ≥90 mL/min).

Group 4 (optional): Participants with moderate renal impairment (eGFR ≥ 30 to < 60 mL/min).

Initially, participants with severe renal impairment (Group 1) and ESRD (Group 2) will be enrolled, along with matching participants with normal renalfunction. An analysis of PK datamay be conducted to determine study progression. The decision to trigger the PK analysis and/or proceed with an evaluation of participants with moderate renal impairment (Group 4) will be made by the sponsor.

Each matched participant with normal renal function (Group 3) enrolled in the study will be demographically matched by sex, age (±10 years), and BMI (±20% kg/m2; data obtained at screening) to an enrolled renal impairment participant. Participants with normal renal function cannot be matched to more than one renally impaired participant within an impairment group; however, participants with normal renal function may be matched to 1 participant from more than 1 renal impairment group.

Potential participants will be screened to assess their eligibility to enter the study up to 4 weeks prior to administration of study intervention. Eligible participants will be admitted to the study site on Day -1. On Day 1, a "A" single oral dose of AZD0780 will be administered, and participants will be confined to the study site until after assessments are completed on Day 11.

For participants with ESRD (Group 2), the first post dose HD session should be scheduled to start 26 hours after administration of AZD0780. Subsequent HD sessions should be scheduled as clinically appropriate.

Serial PK (venous) blood samples will be collected up to 240 hours postdose and urine samples will be collected up to 96 hours postdose for the measurement of AZD0780. Urine collection is not required for participants who are anuric (ie, participants with ESRD on HD [Group 2]). For participants with ESRD (Group 2), blood samples for PK analysis will also be collected prior to, during, and at the end of HD. The entire dialysate will be collected in separate hourly collections on Day 2 for participants with ESRD (Group 2) for the measurement of AZD0780. The volume of each hourly collection of dialysate from which a sample is taken will be recorded. Physical examinations, 12-lead electrocardiograms, vital sign measurements, and clinical laboratory tests will be performed to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

- Participant must be 18 to 85 years of age, inclusive at the time of signing ICF

For Participants with normal renal function:

- Participant must be medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, or 12-lead ECGs, as deemed by the investigator at screening and Day -1

For Participants with renal impairment:

* Diagnosis of chronic kidney disease, stable renal function in the 6 months prior to dosing
* Received HD for chronic renal failure for at least 3 months prior to dosing (Group 2)
* Participants with renal impairment, as follows, based on CKD-EPI equation (BSA-adjusted eGFR) at screening: Group1 eGFR < 30 mL/min), not requiring dialysis, Group 2 ESRD (eGFR < 15 mL/min) on a stable intermittent HD schedule for at least 3 months prior to planned dosing and Group 4 (optional) moderate renal impairment (eGFR ≥ 30 to < 60 mL/min)
* Male participants:
* Males must be surgically sterile or using, in conjunction with their female partner, a highly effective method of contraception for the duration of the study (from the time of study intervention administration) until 3 months after discharge to prevent pregnancy in a partner.
* Female participants of non-childbearing potential:
* Female participants must not be pregnant and must have a negative pregnancy test at screening and check-in, must not be lactating, and must not be of childbearing potential.

Exclusion Criteria:

For Participants with normal renal function:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment).
* Use of any prescription or non-prescription drugs (including vitamins, recreational drugs, and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before study intervention, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* History of any major surgical procedure within 30 days prior to study intervention.

For Participants with renal impairment:

* Presence of unstable medical or psychological conditions which, in the opinion of the investigator, would compromise the participant's safety or successful participation in this study.
* Renal transplant patients (participants on HD with non-functioning renal transplants are not excluded), participants waiting for organ transplant scheduled to occur during the study, and those with a history of acute kidney injury occurring within 3 months prior to screening.
* History of any major surgical procedure within 30 days prior to study intervention.
* Current or previous treatment with drugs for reduction or inhibition of PCSK9 (eg, evolocumab, alirocumab, or inclisiran).
* Use of moderate/strong inhibitors or inducers of CYP3A4/5.
* Unable to refrain from potassium binders, phosphate binders (eg, aluminium hydroxide and calcium carbonate), cholestyramine/colestipol, and ranitidine/nizatidine within 10 hours before and 10 hours after study intervention.
* Receiving or has received within 14 days of screening, medication that contains a black box warning for significant QT prolongation. A list of prohibited medications can be found in protocol.
* Use of concurrent medication which affects calculation of eGFR by affecting serum creatinine (eg, cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine, or quinine) within 7 days of Day -1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
AUClast | From Day 1 to Day 11
  Area under the concentration-time curve from zero to the last measurable concentration
Cmax | From Day 1 to Day 11
  Maximum observed plasma concentration
AUCinf | From Day 1 to Day 11
  Area under the concentration-time curve from zero to infinity

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From Day 1 to Day 11
  To assess the safety and tolerability of a single oral "A" dose for participants with severe renal impairment (not on dialysis), ESRD on HD, and moderate renal impairment (optional) and those with normal renal function
Number of participants with abnormal vital signs, abnormal ECGs, and abnormal physical examination findings | From Day 1 to Day 11
  To assess the safety and tolerability of a single oral "A" dose for participants with severe renal impairment (not on dialysis), ESRD on HD, and moderate renal impairment (optional) and those with normal renal function
Number of participants with abnormal laboratory test results | From Day 1 to Day 11
  To assess the safety and tolerability of a single oral "A" dose for participants with severe renal impairment (not on dialysis), ESRD on HD, and moderate renal impairment (optional) and those with normal renal function
PK parameters Tmax | From Day 1 to Day 11
  Time to reach maximum observed plasma concentration
PK parameters t1/2λz | From Day 1 to Day 11
  half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve
PK parameters CL/F | From Day 1 to Day 11
  apparent total body clearance of drug from plasma after extravascular administration
PK parameters CLNR/F | From Day 1 to Day 11
  Non-renal clearance of drug from plasma after oral administration
PK parameters Vz/F | From Day 1 to Day 11
  Apparent volume of distribution during the terminal phase after extravascular administration
PK parameters AUC0-96 | From Day 1 to Day 11
  area under the concentration-time curve from zero to 96 hours postdose
PK parameters CLr | From Day 1 to Day 11
  renal clearance of the drug from plasma
PK parameters Ae | From Day 1 to Day 11
  cumulative amount of unchanged drug excreted into the urine
PK parameters Fe | From Day 1 to Day 11
  Fraction of the drug excreted into the urine

CONTACTS AND LOCATIONS:
Overall Officials: Kwabena Ayesu, Medicine, Principal Investigator — Omega Research Orlando; Thomas Marbury, Medicine, Principal Investigator — Orlando Clinical Research Center; Juan Carlos Rondon, Medicine, Principal Investigator — Clinical Pharmacology of Miami, Inc.; Trisha Shamp, Medicine, Principal Investigator — Nucleus Network; Joel Neutel, Medicine, Principal Investigator — Orange County Research Center
Locations (4):
- United States (4):
  - Research Site, Lake Forest, California
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida
  - Research Site, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/